CLINICAL TRIAL: NCT07209306
Title: Testing the Effectiveness and Implementability of WHO Psychological Intervention Strategies for Improving Mental Health Outcomes in Migrant Populations Resettled in Italy: the ADVANCE Randomized Controlled Trial
Brief Title: WHO Psychological Interventions for Mental Health Outcomes in Migrants Resettled in Italy: the ADVANCE Trial
Acronym: ADVANCE-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Corrado Barbui, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 101080323; European Commission (Other Grant/Funding Number: Horizon EU Grant Agreement 101080323)
Record Dates: First submitted 2025-09-10; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Distress, Psychological; Distress, Emotional
Keywords: Migrant populations; Psychological distress; Psychological wellbeing; WHO psychological interventions; Effectiveness; Implementation; Self-Help Plus; Doing What Matters in Times of Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be assessed by a trained masked assessor. Secondary outcomes will be self-assessed through validated rating scales. Moreover, the statistical analysis will be masked, i.e., we will use coded groups for the trial statistician for the ITT analysis. Moreover, the trial statistician will not be involved in determining participants' eligibility, in administering the intervention, in measuring the outcomes or in entering data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Help Plus and booster session (Experimental): SH+ program, composed of 5 sessions, and a booster session.
  All participants in the three arms will receive WHO PFA and ECAU, that will include an information flyer about locally available services for migrants.
  Interventions: Other: Experimental: Self-Help Plus and booster session
- Doing What Matters in Times of Stress and booster session (Experimental): DWM and booster session. All participants in the three arms will receive WHO PFA and ECAU, that will include an information flyer about locally available services for migrants.
  Interventions: Other: Doing What Matters in Times of Stress and booster session
- Psychological placebo (Placebo Comparator): Psychological placebo will consist of a phone call or online meetings with a helper, of the same duration of the DWM sessions.
  Additional session: The additional session of psychological placebo will be provided individually in an online format. It will contain neutral contents and will be facilitated by a helper. It will have the same duration as the booster sessions.
  Interventions: Other: Psychological Placebo

INTERVENTIONS:
Other: Experimental: Self-Help Plus and booster session — The SH+ programme, developed by WHO is a five-session stress management course. Supervised non-specialist facilitators will deliver it in a group setting in person. SH+ is intended to be transdiagnostic, easily adaptable to different cultures and languages and both meaningful and safe for people with and without mental disorders.
  Booster session:
  The booster session of SH+ will be provided individually to participants in an online format. It will last approximately 45 minutes, and it will contain a summary of the main contents of the five sessions. The booster session has been developed according to WHO manuals and will be delivered by a trained facilitator.
  All participants in the three arms will receive ECAU that will include an information flyer about locally available services for migrants (education, health, social and legal support), and may include community care, social/legal support, etc.
  Arms: Self-Help Plus and booster session
Other: Doing What Matters in Times of Stress and booster session — Arm Description: The DWM program has been developed by WHO as a stress management guide for coping with adversity. DWM contains the same content as the SH+ illustrated guide, training the five basic stress management skills with standalone audio. Additionally, participants are guided by a briefly trained helper. In this study, the DWM program will be delivered individually as an online guided intervention. The DWM intervention has been adapted for use on a smartphone or other device with internet access. In the online application tool, a new module (i.e., section) is released every week so participants will be asked to go through the entire DWM intervention within five weeks, with guidance from a helper through brief we brief weekly phone or text-based contacts of approximately 15 minutes. Booster session: The booster session will be provided online individually. It has been developed according to the WHO manual, and it contains a summary of the main contents of the online sessions.
  Arms: Doing What Matters in Times of Stress and booster session
Other: Psychological Placebo — Psychological placebo will consist of a phone call or online meetings with a helper, of the same duration of the DWM sessions. In the first part of the call participants will be reminded about locally available social, health, legal and education services. In the second part of the call participants will choose a discussion topic from topics presented in a list prepared by the research team . Additional session: The additional session of psychological placebo will be provided individually in an online format. It will contain neutral contents and will be facilitated by a helper. It will have the same duration as the booster sessions.
  Arms: Psychological placebo

SUMMARY:
Rationale: Migrant populations face numerous mental health risk factors, including unmet expectations, inadequate support, acculturation challenges, and legal hurdles. These stressors hinder their lives during and after migration. The World Health Organization has developed scalable psychological interventions, including Self Help Plus (SH+) and its online version Doing What Matters in Times of Stress (DWM), which are designed for delivery by non-professional helpers and adaptable to various cultures and mental health issues. While initial randomized controlled trials (RCTs) show these interventions are effective, their medium to long-term efficacy, implementability and scalability have not been thoroughly evaluated.

Objectives: This study aims to examine the efficacy of SH+ and DWM versus a psychological placebo in reducing anxiety and depression symptoms among migrants experiencing elevated psychological distress. Additionally, it seeks to collect implementation outcomes to assess the feasibility and potential for scaling up these interventions.

Study design: We will conduct a hybrid three-arm efficacy-implementation randomized controlled trial.

Study population Adult asylum seekers, refugees or migrants with self-reported elevated psychological distress (K10 >15.9) (n=237).

Intervention : All participants (in the three comparison groups) will receive Psychological First Aid (PFA) and enhanced care as usual (ECAU). In addition to PFA and ECAU, the intervention group 1 will receive SH+ complemented with an online booster session (delivered 4 weeks after SH+), the intervention group 2 will receive DWM complemented with an online booster session (delivered 4 weeks after DWM), and the intervention group 3 will receive psychological placebo (PsychP) complemented with an online session with neutral contents of the same duration of groups 1 and 2 (delivered 4 weeks after PsychP).

Main study parameters/endpoints: Screening for inclusion and exclusion criteria will be interviewer-administered, in-person or through (video) calls. For all participants, online assessments will take place at baseline, at 4/6 weeks after having received DWM (which corresponds to 1 week after the booster session, and 3 months after randomization), and at 6 months after randomization. The primary outcome will be the decrease in symptoms of anxiety and depression from baseline to three-month after randomization, measured through the sum score of the Patient Health Questionnaire (PHQ-9) and General Anxiety Disorder-7 (GAD-7), i.e. the PHQ-Anxiety and Depression Score (PHQ-ADS). We expect to detect a Cohen's d effect size of 0.3 in the SH+ and DWM groups at 3 months after randomization. Additional health outcomes include level of anxiety (GAD-7) and depression (PHQ-9), functional impairment (WHODAS), wellbeing (WHO-5), quality of life (EQ-5D-5L), and cost of care (CSRI). Implementation outcomes will be measured with the Adoption of Information, Technology measure, Measure of Disseminability and Levels of Institutionalization tool, adverse events, and WHO fidelity forms. Additional study parameters include demographic data and dropouts.

DETAILED DESCRIPTION:
The World Health Organization (WHO) has developed a number of scalable psychological interventions for populations affected by adversity. These include Self Help Plus (SH+) and its online version Doing What Matters in Times of Stress (DWM). A core feature of all WHO scalable interventions is that they can be delivered by non-professional helpers, such as a trained peer, or helper at the workplace, or a psychosocial worker after receiving training (task-shifting). The interventions have been designed to be widely applicable to a variety of mental health conditions, such as depression, anxiety and PTSD, and easily adaptable to different populations, cultures and languages. Additionally, the interventions and their implementation materials are open access and available on the WHO website. SH+ builds on existing innovations in delivery of mental health interventions for vulnerable population groups, and focuses on psychological distress broadly, by teaching stress management skills that might be applied across a range of difficulties. It has been implemented with different populations of asylum seekers and refugees in Europe, Turkey and Northern Uganda. The online version of SH+ is called "Doing What Matters in Times of Stress" (DWM). DWM was originally designed for flexible implementation either in a group or individual format throughout a digital format. In the guided version of DWM, participants also receive support from a trained helper. DWM is based on Acceptance and Commitment therapy (ACT), a modern form of cognitive-behavioral therapy with a strong focus on mindfulness practices and includes exercises which aim to enhance stress reduction and build social support, adaptive coping and resilience. People can use the self-help intervention in their own time. The intervention consists of five weekly sessions which follow the five chapters of the SH+ book (grounding, unhooking, acting on your values, being kind and making room). Participants receive a weekly call from a so-called "helper" to support them accessing the intervention sessions, and to provide guidance in using the skills in everyday life.

The DWM version of SH+ has been tested in three RCTs focused on vulnerable populations (i.e., migrants and people in social adversity) in Europe and in one RCT involving health workers in Spain as part of the RESPOND project, and in a RCT with health workers during the COVID-19 pandemic in Italy.

Although data from RCTs indicate that these intervention strategies are initially effective, their efficacy appears to diminish over the medium to long term. Furthermore, the feasibility and potential for scaling up these interventions have not yet been formally evaluated in implementation studies.

Against this background, the present study aims to examine the efficacy of SH+ and DWM versus psychological placebo in reducing anxiety and depression symptoms in a group of migrants experiencing elevated psychological distress. Additionally, the study seeks to collect implementation outcomes to assess the feasibility and potential for scaling up these interventions.

OBJECTIVES:

Primary objective: The primary aim of this RCT is to evaluate the efficacy and implementability of three intervention strategies:

1. The culturally and contextually adapted WHO intervention programme SH+, delivered in groups of up to 20 people, in person, and complemented with a booster session;
2. The culturally and contextually adapted WHO intervention programme DWM, delivered as a guided online individual intervention, and complemented with a booster session;
3. A psychological placebo condition, administered online individually with the same frequency and dosage of the WHO intervention programmes, and consisting of phone calls or online meetings with a helper.

   This evaluation specifically targets the adult migrant population resettled in Italy, focusing on the reduction of psychological distress.

   Secondary objective: the secondary objective of this trial is to conduct a comprehensive economic evaluation to assess the economic costs, cost-effectiveness, extended cost-effectiveness, and budget impact of implementing the two aforementioned interventions (SH+ with a booster session and DWM with a booster session) compared to the psychological placebo condition. The cost-effectiveness will relate the costs to the health effects of delivering the two interventions in relation to the psychological placebo condition to determine whether the interventions present a more efficient use of resources. Additionally, the extended cost-effectiveness analysis will relate costs to the non-health effects of the interventions (e.g. improvement of financial health protection measured as reduction in out-of-pocket expenditure for care services) and examines the intervention effects on equity by quantifying how the effects are distributed across different socio-economic groups. The findings of the economic evaluation are expected to inform the decisions on adoption and scaling up of SH+ and DWM for the prevention and promotion of mental health among the migrant population in Italy and similar European countries.

   STUDY DESIGN: This is a hybrid efficacy-implementation RCT comparing different implementation strategies of WHO psychosocial interventions against a psychological placebo. The study will compare the SH+ intervention with a booster session, the DWM with a booster session, and psychological placebo. Participants will be adult migrants (> 18 years) screened for elevated psychological distress (Kessler Psychological Distress Scale > 15.9) resettled in Italy. Before random allocation, all participants eligible for inclusion will receive Psychological First Aid according to the WHO protocol. Then, participants will be randomly allocated to receive SH+ with a booster session (intervention group 1), DWM with a booster session (Intervention group 2), or psychological placebo with an online additional session (intervention group 3).

   All participants will also receive enhanced care as usual (ECAU) consisting of information materials (i.e., flyers) about locally available referral options, and social and legal services for migrant population groups resettled in Italy.

   STUDY POPULATION: Population: Participants will be adult migrants (> 18 years) resettled in Italy. Recruitment will be conducted in Verona and Rome. Participants will be recruited through (a) local organizations, including governmental and non-governmental organizations (NGOs), (b) target social media recruitment (e.g., Facebook, Instagram, TikTok), and word of mouth, (c) other community-based organizations offering legal, social, administrative, psychological, or religious support for this vulnerable group.

   Inclusion criteria: Participants will be eligible to participate in the study if they meet the following criteria:
   * 18 years or older
   * Living in Italy temporarily or permanently as a migrant, including asylum seekers, refugees, labor migrants ((IOM), 2019);
   * Having elevated levels of psychological distress (K10 >15.9);
   * Sufficient mastery (written and spoken) of one of the languages the SH+/DWM intervention is being delivered in (i.e., English and/or Italian);
   * Oral and written informed consent before entering the study.

   Exclusion criteria: Potential participants who meet the inclusion criteria will be excluded from participation in this study if they meet any of the following criteria:
   * Planning to permanently move back to their home country before the last follow-up assessment (at six months after randomization);
   * Having acute medical conditions (requiring hospitalization);
   * Imminent suicide risk, or expressed acute needs or protection risks that require immediate follow-up based on screening tool and clinical judgement;
   * Having a severe mental disorder (e.g., psychotic disorders, substance-dependence) based on clinical judgement;
   * Having severe cognitive impairment based on clinical judgement (e.g., severe intellectual disability or dementia);
   * Currently receiving specialized psychological treatment (e.g., Cognitive Behavioral treatment (CBT), Eye Movement Desensitizing and Reprocessing (EMDR));
   * In case of current psychotropic medication use: being on an unstable dose for at least two months.

   Sample size calculation: A total number of 237 participants will be included. Based on findings from previous SH+ studies, a Cohen's f effect size of .34 for the time-by-treatment interaction at post-intervention is hypothesized between each active arm (SH+ and DWM) and the psychological placebo arm at 3 months post randomization based on the primary outcome PHQ-ADS. The PHQ-ADS is the combined sum score of depression and anxiety symptoms of the PHQ-9 and GAD-7 respectively and has shown good internal consistency (α = .88 to .92).

   The Benjamini-Hochberg correction for multiplicity will be applied. Power calculations for the ANOVA within-between interaction are based on the case of lack of significance of the other intervention, thus a p-value of 0.025 was considered. To guarantee a 90% power for each test, 55 participants per study arm will be required. Finally, to take a 30% attrition into account, 79 participants per arm will be needed, thus a 3-armed RCT with 237 participants will be conducted.

   INTERVENTIONS:

   Psychological First Aid (PFA) (All participants):

   Before randomization, all eligible participants will be offered individual Psychological First Aid (PFA) through a face-to-face or teleconferencing meeting. PFA is a WHO developed support strategy that involves humane, supportive, and practical help for individuals suffering from serious humanitarian crises. PFA does not necessarily involve a discussion of the event(s) that cause the distress but aims particularly at five basic elements that are crucial to promote in the aftermath of crises, i.e., a sense of safety, calm, self- and community efficacy, connectedness, and hope. PFA consists of a (telephone) conversation (approximately 30-45 minutes) that a helper has with a participant. The helper provides non-intruding practical care and support, assesses needs and concerns, helps people to address basic needs (e.g., information), listens to people without pressuring them to talk, comforts people and helps them to feel calm, helps people to connect to information, services and social support, and protects people from further harm.

   Enhanced Care-as-usual (ECAU) (All participants):

   In addition to PFA, all participants in the three arms will receive Enhanced Care As Usual (ECAU) that will include an information flyer about locally available services for migrants (education, health, social and legal support), and may include community care, social/legal support, and psychoeducation.

   Because migrants may have a lack of knowledge of the Italian health care system and therefore may not utilize health care, flyers will be distributed to provide information about the Italian health care system and locally available referral options. For all participants, information on whether they have a general practitioner will be collected, provided consent for this recording is obtained. In case the participant gives approval, name and contact details will be recorded.

   Self Help Plus (SH+) (Intervention arm 1):

   The SH+ programme, developed by WHO and humanitarian collaborators, is a five-session stress management course. Supervised non-specialist facilitators will deliver it in a group setting in person. SH+ was designed to be relevant for large segments of adversity-affected populations: it is intended to be transdiagnostic, easily adaptable to different cultures and languages and both meaningful and safe for people with and without mental disorders.

   Based on Acceptance and Commitment Therapy (ACT), a form of Cognitive-Behavioral Therapy (CBT), SH+ emphasized the concept that ongoing attempts to suppress unwanted thoughts and feelings can paradoxically make these problems worse. Instead, it highlights learning new ways to accommodate difficult thoughts and feelings, while guiding people to take proactive steps towards living in a way that is consistent with their values. ACT has been shown to be useful for a range of mental health issues and has been used successfully in a guided self-help format.

   Therefore, SH+ includes ACT techniques that aim to help people cope with stress, respond compassionately to themselves and others and to live in accordance with their values. The SH+ programme has two components: a pre-recorded course and an illustrated self-help book. Pre-recorded audio material is delivered across five two-hour sessions (or modules) to groups of up to 30 people. The audio material imparts key information about stress management and guides participants through individual exercises and small group discussions. To augment the audio recordings, the illustrated self-help book reviews all essential content and concepts. Written manuals help non-specialist facilitators to conduct the course using the pre-recorded audio.

   The potential value of using a psychoeducational course to access hard-to-reach populations has been shown previously. Evidence for the use of books in interventions is also promising. Furthermore, research has found that guided self-help programmes produce much better results than 'pure' self-help, and the effects produced are like face-to-face psychological treatment (mhGAP, 2010). Furthermore, randomized controlled trials have shown that SH+ has proven effective in promoting mental health prevention among refugee and asylum seeker populations in Western Europe (including Italy) and Turkey.

   Booster session:

   The booster session of SH+ will be provided individually to participants in an online format. It will last approximately 45 minutes, and it will contain a summary of the main contents of the five sessions. The booster session has been developed according to WHO manuals and will be delivered by a trained facilitator.

   Protocol adherence:

   Adherence to the SH+ protocol will be assessed using WHO ad-hoc forms completed by the facilitators. Additionally, the intervention supervisor (a clinical psychologist or a psychiatrist) will observe at least 10% of the sessions completing an adherence form.

   Doing What Matters in Times of Stress (DWM) (Intervention arm 2):

   The DWM program has been developed by WHO as a stress management guide for coping with adversity. Based on ACT, DWM contains the same content as the SH+ illustrated guide, training the five basic stress management skills with standalone audio. Additionally, participants are guided by a briefly trained helper.

   In this study, the DWM program will be delivered individually as an online guided intervention. The DWM intervention, i.e., both the audios and the self-help guide, have been adapted for use on a smartphone or other device with internet access. The format of DWM is innovative in that it seeks to ensure that key intervention components are delivered as intended using pre-recorded audio, without the burden of extensive training and supervision. In the online application tool, a new module (i.e., section) is released every week so participants will be asked to go through the entire DWM intervention within five weeks, with guidance from a helper through brief weekly phone or text-based contacts of approximately 15 minutes. Due to its format, the DWM program does not require much time from experts for implementation. The delivery mode for the support from the helper will be flexible.

   The DWM in its digital format has previously been tested with the same target population (i.e., migrants) in other RCTs, showing promising results in preventing common mental health conditions and promoting psychological well-being.

   Booster session: The booster session of DWM will be provided individually in an online format. It has been developed according to the WHO manual, and it contains a summary of the main contents of the online sessions. The booster session will be facilitated by a trained helper.

   Protocol adherence:

   Adherence to the DWM protocol will be assessed at post-intervention based on meta-data collected during the intervention (i.e., by tracking participants usage of the DWM app, such as who accesses what page, how often, how much time participants spend on the app etc.). This meta-data will be used during the intervention to remind each participant (e.g., through e-mail) after finishing each module to let them know that they should start a new module. Moreover, participants will receive a weekly phone call from a helper to see how they are doing and to check on their progress. Finally, the intervention supervisor (a clinical psychologist or a psychiatrist) will observe at least 10% of the phone contacts.

   Psychological placebo (intervention arm 3):

   Psychological placebo will consist of a phone call or online meetings with a helper, of the same duration of the DWM sessions. In the first part of the call participants will be reminded about locally available social, health, legal and education services. In the second part of the call participants will choose a discussion topic from topics presented in a list prepared by the research team.

   Additional session: The additional session of psychological placebo will be provided individually in an online format. It will contain neutral contents and will be facilitated by a helper. It will have the same duration as the booster sessions.

   Training:

   The personnel delivering the interventions will receive appropriate training and supervision according to the WHO protocols.

   Randomization:

   After the screening and the baseline assessment, participants will receive WHO PFA and will then be randomized to intervention group 1 (SH+) (n= 79), intervention group 2 (DWM) (n = 79) or intervention group 3 (PsychP)(n = 79), with an equal probability of assignment to each group (allocation ratio 1:1:1).

   The randomization will be stratified according to the recruiting site (Verona or Rome) and carried out through computerized software (e.g., REDCap) using permuted block size (e.g., 6-12 participants per block) and will be performed by an independent person who is not involved in the intervention delivery or assessment of participants. Participants randomized to intervention group 1 will be allocated to an SH+ helper, those in intervention group 2 to a DWM helper, those to intervention group 3 to a psychological placebo helper. The allocated helper will send an e-mail to the participant to set up a time and date for a first acquaintance telephone call before the intervention starts.

   Statistical analysis:

   The statistical analysis of the RCT will estimate the efficacy of the intervention programmes SH+ with booster session and DWM with booster session compared with psychological placebo with a neutral additional session. The PHQ-ADS score at three months post-randomization is the primary study outcome. The primary outcome will be summarized using number of subjects (n), minimum and maximum; and means, standard deviations (SD) for normally distributed data, or medians and inter-quartile ranges for non-normally distributed data. To compare at baseline the two intervention groups, standardized mean differences (SMDs) will be calculated. In addition, a covariate-adjusted mixed model of primary outcome will be performed by adding covariates showing imbalance at baseline (as measured by a Standardized Mean Difference above 0.1 in absolute value).

   Both intention-to-treat (ITT) analysis, including all randomized participants (n=237), and completers' (per protocol - PP) analysis will be carried out. The main conclusion of the trial will be based on the ITT analysis of the primary outcome. A secondary analysis of the primary outcome will also be presented using the PP population.

   The statistical analysis will be masked, i.e., we will use coded groups for the trial statistician for the ITT analysis. Moreover, the trial statistician will not be involved in determining participants' eligibility, in administering the intervention, in measuring the outcomes or in entering data. To estimate the treatment effect, a linear mixed model will be employed for the primary endpoint analysis, which will have treatment as fixed effects, baseline measurement of primary endpoint as covariate, and subject as random effects. The mean difference between the study arms at each visit/time together with its 95% confidence interval will be derived from the mixed model. Covariate-adjusted mixed model of primary endpoint will also be performed by adding pre-specified covariates at baseline (gender, age, education, country of origin) into the above model.

   Missing data:

   Missing data will be treated as missing at random (MAR). No imputations of missing values will be made, as multilevel models can deal with missing data at the outcome level.

   Secondary outcome(s):

   Secondary outcomes will be analyzed using repeated measurements. Additionally, a linear mixed model as mentioned for the primary outcome analysis (PHQ-ADS) will be carried out for analysing the following clinical outcomes measured at baseline, at three months post randomization and at six months post randomization: psychological distress (GHQ-12), depressive symptoms (PHQ-9), anxiety symptoms (GAD-7), functioning (WHODAS) and wellbeing (WHO-5).

   Cost-effectiveness analysis:

   Economic evaluation will be conducted from the societal perspective and consists of four sub-components: (1) an activity-based micro-costing study, (2) a cost-effectiveness analysis, (3) a cost-utility analysis, and (4) an extended cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Living in Italy temporarily or permanently as a migrant, including asylum seekers, refugees, labor migrants;
* Having elevated levels of psychological distress (K10 >15.9);
* Sufficient mastery (written and spoken) of one of the languages the SH+/DWM intervention is being delivered in (i.e., English and/or Italian);
* Oral and written informed consent before entering the study.

Exclusion Criteria:

* Planning to permanently move back to their home country before the last follow-up assessment (at six months after randomization);

  * Having acute medical conditions (requiring hospitalization);
  * Imminent suicide risk, or expressed acute needs or protection risks that require immediate follow-up based on screening tool and clinical judgement;
  * Having a severe mental disorder (e.g., psychotic disorders, substance-dependence) based on clinical judgement;
  * Having severe cognitive impairment based on clinical judgement (e.g., severe intellectual disability or dementia);
  * Currently receiving specialized psychological treatment (e.g., Cognitive Behavioral treatment (CBT), Eye Movement Desensitizing and Reprocessing (EMDR));
  * In case of current psychotropic medication use: being on an unstable dose for at least two months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
PHQ-ADS at T2 | T2: 3 months after randomization (1 week after the booster session)
  The primary endpoint will be the symptoms of depression and anxiety measured with the PHQ-ADS scale administered by a masked trained assessor.

SECONDARY OUTCOMES:
PHQ-ADS at T3 | T3: 6 months after randomization (3 months after the booster session)
  Symptoms of depression and anxiety measured with the PHQ-ADS scale
PHQ-9 at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Depressive symptoms measured using the Patient Health Questionnaire depressive module. It asks how often someone was bothered by each of the nine DSM-5 criteria and scores answers on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).
GAD-7 at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Anxiety symptoms assessed with the Generalized Anxiety Disorder 7-item rating scale (GAD-7). The GAD-7 is a self-rated questionnaire consisting of seven items that investigate the level of anxiety and worry experienced by the respondent . Each item is scored on a 0-3 scale, with a total score ranging from 0 to 21. Higher scores indicate more anxiety symptoms during the past two weeks.
GHQ-12 at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Psychological distress measured using the 12-item General Health Questionnaire (GHQ-12) (Goldberg). The GHQ-12 is a measure of current mental health andasks whether the respondent has experienced a particular symptom or behavior recently.
WHODAS at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Functional impairment assessed with the WHO Disability Assessment Schedule 2.0 (WHODAS) interviewer-administered version. The WHODAS is a generic assessment instrument assessing health and disability. It is used across all diseases, including mental, neurological and substance use disorders. We will use the 12-item interviewer-administered version.
WHO-5 at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Subjective wellbeing assessed with the WHO-5 Wellbeing Index (WHO-5) that is a 5-item questionnaire measuring current psychological wellbeing and quality of life. Scores range from 0 to 25.
CSRI at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  The Client Service Receipt Inventory (CSRI) for the collection of data on care service utilization (e.g., use of health care services, social care, time out of employment and other usual activities, need for informal care) and related socio-demographic characteristics of people with mental disorders, as the basis for calculating the costs of care for mental health.
EQ 5D 5L at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  The intervention effects on the health-related quality of life measured as Quality-Adjusted Life Year (QALY) will rely on the use of the EQ-5D-5L, which consists of two main sections: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system encompasses five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension presents five levels of severity: no problems, slight problems, moderate problems, severe problems and extreme problems.
ISMI at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  ISMI, Internalized Stigma of Mental Illness
Implementation outcomes at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Implementation outcomes: fidelity (assessed using WHO fidelity forms and meta-data), acceptability, adoption, feasibility, penetration, and adverse events.
  Adverse events are defined as any undesirable experience occurring to a subject during the study, whether considered related to the trial procedure or the SH+ / DWM intervention. All adverse events reported spontaneously by the subject or observed by the investigator or by the staff will be recorded.
Acceptability of intervention measure (AIM) at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Implementation outcomes: Acceptability, assessed with the "Acceptability of Intervention Measure" (AIM) subscale (4 item, 5-point Likert scale: 1 = completely disagree to 5 = completely agree) (Weiner et al., 2017). The unit of measure is a descriptive scale rating the level of acceptability of the intervention.
Intervention appropriateness measure (IAM) at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Implementation outcomes: Appropriateness, assessed with the "Intervention Appropriateness Measure" (IAM) subscale (4 item, 5-point Likert scale: 1 = completely disagree to 5 = completely agree) (Weiner et al., 2017). The unit of measure is a descriptive scale rating the level of appropriateness of the intervention.
Feasibility of intervention measure (FIM) at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  Implementation outcomes: Feasibility, assessed with the "Feasibility of Intervention Measure" (FIM) subscale (4 item, 5-point Likert scale: 1 = completely disagree to 5 = completely agree) (Weiner et al., 2017). The unit of measure is a descriptive scale rating the level of feasibility of the intervention.
Drop-outs at T2 and T3 | T2: 3 months after randomization (1 week after the booster session) T3: 6 months after randomization (3 months after the booster session)
  The number of participants dropping out from the study and the reason.

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Barbui, MD, Full professor, Principal Investigator — Universita di Verona
Locations (1):
- WHO Collaborating Centre for Research and Training in Mental Health and Service Evaluation Department of Neurosciences, Biomedicine and Movement Sciences, Section of Psychiatry, University of Verona, Verona, Italy., Verona, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be shared upon motivated request and after discussion with the ADVANCE project General Assembly.
Supporting Information: Study Protocol, SAP